CLINICAL TRIAL: NCT02428764
Title: A Multicenter Phase II Trial of Induction Nimotuzumab Plus Gemcitabine and Carboplatin Followed by Surgery in Patients With Unresectable Stage III Squamous Cell Lung Carcinoma
Brief Title: Neoadjuvant Nimotuzumab Plus Gemcitabine and Carboplatin in Unresectable Stage III Squamous Cell Lung Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1010; wsy006 (Other: Guangdong Province Association Study of Thoracic Oncology)
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — nimotuzumab; Gemcitabine; Carboplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention group (Experimental): Patients were assigned to receive neoadjuvant nimotuzumab plus gemcitabine and carboplatin followed by surgery.
  Interventions: Drug: Nimotuzumab; Drug: Gemcitabine; Drug: Carboplatin; Procedure: Surgery

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab was given 200 mg i.v. injection over 30 min on days 1 and 8
Drug: Gemcitabine — Gemcitabine was given 1000 mg/m2 i.v. injection on days1 and 8.
  Other Names: Gemzar
Drug: Carboplatin — carboplatin was given dosed to an area under the serum concentration-time curve (AUC) of 5 i.v. on day 1.
  Other Names: CBP
Procedure: Surgery — Patients' resectability was assessed by a medical team, including thoracic surgeons, medical oncologists, and radiologists.

SUMMARY:
The purpose of this study is studying induction nimotuzumab plus gemcitabine and carboplatin followed by surgery to see how well it works in treating patients with unresectable stage III squamous cell lung carcinoma.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy is the recommended therapeutic approach for patients with unresectable stage III non-small cell lung cancer (NSCLC), although surgery offers the chance of cure. With combined-modality therapy with radiation therapy and chemotherapy, the prognosis of stage III NSCLC remains poor. Nimotuzumab, a human anti-EGFR monoclonal antibody, has shown its efficacy in the treatment of head/neck squamous cell carcinoma, nasopharyngeal carcinoma as well as lung cancer. This study is studying neoadjuvant nimotuzumab plus gemcitabine and carboplatin followed by surgery to see how well it works in treating patients with unresectable stage III squamous cell lung carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Target population is unresectable stage III squamous cell lung carcinoma.
* Written informed consent provided.
* Male and female patients aged ≥18 years, ≤75 years.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy ≥12 weeks.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
* Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min.
* Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Known severe hypersensitivity to nimotuzumab or any of the excipients of this product.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease.
* Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
* Patients with prior chemotherapy or therapy with systemic anti-tumour therapy (e.g. monoclonal antibody therapy).
* Patients with prior radiotherapy
* History of another malignancy in the last 5 years with the exception of the following: other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted. Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or puts the subject at high risk for treatment-related complications.
* Patient who has active serious infection (e.g. pyrexia of or 38.0℃ over).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04-01; Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Resectability rate | 3 months

SECONDARY OUTCOMES:
Number of participants with perioperative complications | 1 year
Event-free survival | 2 years after the last patient is enrolled
  Event-free survival was assessed from diagnosis to disease recurrence/metastasis/progression or death as a result of any cause.
Overall survival | 2 years after the last patient is enrolled
  Overall survival was assessed from diagnosis to death as a result of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Si-Yu Wang, MD, Principal Investigator — Guangdong Province Association Study of Thoracic Oncology
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China